CLINICAL TRIAL: NCT04598269
Title: A Phase 2a, Multicenter, Randomized, Double-blind, Vehicle-controlled, Parallel-group Study to Determine the Safety, Tolerability, Pharmacokinetics and Efficacy of ATI-1777 in Adult Patients With Moderate or Severe Atopic Dermatitis
Brief Title: Study of ATI-1777 in Adult Patients With Moderate or Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATI-1777-AD-201
Record Dates: First submitted 2020-10-05; First posted 2020-10-22 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Vehicle-controlled, Parallel-group Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ATI-1777 (Experimental): ATI-1777 topical solution 2.0% w/w, twice daily
  Interventions: Drug: ATI-1777
- Vehicle (Placebo Comparator): Vehicle topical solution, twice daily
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: ATI-1777 — ATI-1777 topical solution 2.0% w/w
  Arms: ATI-1777
Drug: Vehicle — Vehicle topical solution containing no ATI-1777
  Arms: Vehicle

SUMMARY:
This is a first-in-human, randomized, double-blind, parallel-group, vehicle-controlled study to evaluate the efficacy, safety, tolerability, and PK of ATI-1777 solution following twice-daily applications to target areas of participants with moderate or severe atopic dermatitis (AD).

DETAILED DESCRIPTION:
Participants underwent screening evaluations to determine eligibility up to 30 days prior to randomization. Participants who meet all the entry criteria were randomized on Day 1 to active or vehicle treatment. Participants applied study drug (ATI-1777 topical solution 2.0% w/w or vehicle) twice daily for 4 weeks with weekly study visits and were to return 2 weeks after the last dose of study medication for a Post treatment Follow-up (PTFU) Visit.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign the IRB approved informed consent form (ICF) prior to administration of study-related procedures.
2. Male patients or non-pregnant, non-nursing female patients 18 to 65 years old, inclusive, at the time of informed consent.
3. Pregnancy and Contraception:

   * Women of childbearing potential (WOCBP), must have a negative serum pregnancy test at the Screening Visit, a negative urine pregnancy test immediately prior to the first application of study medication on Day 1, and a negative urine pregnancy test at each study visit thereafter.
   * WOCBP must agree to use 2 forms of highly effective contraception, including 1 physical barrier (condom or diaphragm) plus another highly effective method, such as adequate hormonal method (e.g., contraceptive implants, injectables, oral contraceptives) or nonhormonal methods (e.g., intrauterine device, spermicidals) throughout the Screening Period and until 30 days after the last administration of study medication.
   * Male patients with partners of childbearing potential may be enrolled if they are:

     * Documented to be surgically sterile (vasectomy), or
     * Using 2 adequate forms of highly effective contraception, 1 of which should be a physical barrier until 90 days after the last administration of study medication.
4. Have a diagnosis of AD fulfilling the specified diagnostic criteria of Hanifin and Rajka (Hanifin and Rajka 1980).
5. Have at least a 6-month history of AD prior to the Screening Visit, and no significant AD flares for the 4 weeks prior to the Screening Visit.
6. Have at least 1 lesion that measures at least 3 cm2 at the Screening Visit and on Day 1 prior to the first dose of study medication. This lesion must be representative of the patient's disease state, but not located on the hands, feet, or genitalia.
7. Have a stable diagnosis of moderate or severe (IGA score 3 or 4) AD at the Screening Visit.
8. Have AD affecting 3% to 20% BSA (not including scalp, face, palms of hands, soles of feet, groin, and genitalia) at the Screening Visit.
9. Willing to refrain from washing area of treatment or swimming for 6 hours after each study medication application.
10. Willing to refrain from excessive sun exposure (e.g., sunbathing and/or tanning salon visits) and to minimize sun exposure (e.g., wear sun protective clothing, hat) as much as possible.
11. Willing to refrain from use of moisturizers, emollients, and sunscreen on AD study treatment areas for duration of protocol therapy.
12. Willing to refrain from participating in strenuous exercise that would cause profuse sweating for a period of 6 hours after each study medication application.
13. Willing to return to the clinic, follow all study instructions, attend all study visits, and complete study procedures.
14. In good general health and free of any known disease state or physical condition that, in the investigator's opinion, might impair evaluation of the patient or that might expose the patient to an unacceptable risk by study participation.
15. Willing and capable of taking appropriate coronavirus disease 2019 (COVID-19) risk mitigation precautions (e.g., wearing a mask in public, adhering to social distancing, etc.) as recommended or required by local, state, or federal guidelines during participation in the study.

Exclusion Criteria:

1. Unstable course of AD (spontaneously improving or rapidly deteriorating) based on the patient history or as determined by the investigator during the Screening Period.
2. Refractory AD (i.e., AD that required frequent hospitalizations and/or frequent intravenous treatment for skin infections within the year before the Screening Visit).
3. AD of a severity (EASI >48) that the patient is not a candidate for a vehicle-controlled study.
4. Any signs or symptoms associated with AD therapy (e.g., history of anaphylaxis, hypersensitivity reactions, skin atrophy, striae, pigmentary changes) that, in the investigator's opinion, might impair evaluation of the AD or which exposes the patient to unacceptable risk by study participation.
5. Concomitant skin disease or clinically infected AD or presence of other skin disease in the area to be dosed that may interfere with study assessments.
6. Use of any of the following treatments within the indicated washout period prior to Day 1:

   * Phototherapy (ultraviolet A, ultraviolet B, or psoralen and ultraviolet A therapy) within 4 weeks prior to Day 1.
   * Systemic biologic immunosuppressant or immunomodulatory therapy (e.g., etanercept, alefacept, infliximab, dupilumab) within 12 weeks (or 5 half-lives of the product, whichever is longer) prior to Day 1.
   * Non-biologic immunosuppressants (e.g., methotrexate, retinoids, calcineurin inhibitors, cyclosporine, hydroxycarbamide [hydroxyurea], azathioprine) within 4 weeks prior to Day 1.
   * Janus kinase (JAK) inhibitors (systemic and topical) within 4 weeks prior to Day 1.
   * Systemic corticosteroids within 2 weeks prior to Day 1 (intranasal, inhaled, and topical ocular corticosteroids are allowed).
   * Cytostatic agents within 4 weeks prior to Day 1.
   * Crisaborole within 2 weeks prior to Day 1.
   * Systemic antibiotics within 30 days prior to Day 1.
   * Topical treatments for AD (corticosteroids, calcineurin inhibitors, topical H1 and H2 antihistamines, topical antimicrobials, and other medicated topical agents) within 2 weeks prior to Day 1.
   * Live attenuated vaccine treatment within 12 weeks prior to Day 1.
   * Other investigational product within 30 days or 5 half-lives (whichever is longer) prior to Day 1.
7. Previous failure to respond to prior therapy with JAK inhibitors (systemic or topical), as determined by the investigator.
8. Current use of an oral H1 antihistamine (e.g., diphenhydramine, terfenadine) unless the patient is on a stable dose for at least 14 days prior to the Screening Visit.
9. Medical marijuana unless the patient is on a stable dose for at least 14 days prior to the Screening Visit.
10. Clinically significant laboratory abnormalities at the Screening Visit that, in the opinion of the investigator, could affect interpretation of study data or the safety of the patient's participation in the study.
11. Clinical laboratory values:

    * White blood cell count <2×109/L
    * Absolute neutrophil count (ANC) <1800/mL
    * Platelet count <130,000/mL
    * Hemoglobin <8g/dL
    * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2× the upper limit of normal
    * Lymphocyte count <0.5×109/L
12. Investigator-assessed history of, or current physical findings of, severe, progressive, or uncontrolled immunologic, hepatic, gastrointestinal, pulmonary, cardiovascular, genitourinary (renal), hematological, neurologic or cerebral disorders, infectious disease or coagulation disorders that, as determined by the investigator, could affect the safety of the patient's participation in the study or would preclude participation in and completion of study assessments.
13. History of, current, or suspected systemic or cutaneous malignancy and/or lymphoproliferative disease within the last 5 years, other than patients with a history of adequately treated and well healed and completely cleared nonmelanoma skin cancers (i.e., basal or squamous cell carcinoma) or cervical carcinoma in situ treated successfully at least 1 year prior to the Screening Visit 1 with no evidence of disease.
14. Evidence of active, chronic, or latent infections at the time of enrollment or a systemic infection including but not limited to a history of treated infection (e.g., pneumonia, septicemia) within 3 months prior to Day 1.
15. Patient has a known active or history of incompletely treated or untreated active tuberculosis. Patients with a history of active tuberculosis must have documented adequate treatment verified by the investigator. Patients who demonstrate evidence of latent tuberculosis infection (positive QuantiFERON® Tuberculosis Gold Test) will only be allowed to participate in the study if there is documented evidence of a completed adequate treatment course for latent tuberculosis and if active tuberculosis is excluded per the investigator's judgment.
16. History of a serious local skin infection (e.g., cellulitis, abscess) within 5 years of the Screening Visit.
17. Positive serological test for human immunodeficiency virus (HIV) (antibody), hepatitis C virus (antibody), hepatitis B surface antigen, or hepatitis B core antigen antibody.
18. Known significant exposure (close contact [<6 feet] for ≥15 minutes) to an individual with a confirmed diagnosis of coronavirus disease 2019 (COVID-19) at any time during the Screening Period.
19. Herpes zoster or cytomegalovirus infection that resolved less than 2 months prior to the Screening Visit. Patients with a history of frequent outbreaks of herpes simplex virus (defined as 4 or more outbreaks a year).
20. Clinically significant electrocardiogram (ECG) findings such as, but not limited to, baseline mean QTcF >450 msec for males or >470 msec for females (use of the ECG algorithm is acceptable for this purpose).
21. Known allergy to any of the inactive ingredients in the study drug.
22. Female patients who are pregnant, nursing, or planning to become pregnant during the study.
23. Legal incapacity or limited legal capacity.
24. Major surgery within 3 months of the Screening Visit.
25. Any other condition that precludes adequate understanding, cooperation, and compliance with study procedures or any condition that could pose a risk to the patient's safety, as per the investigator's judgment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Aclaris Investigational Site, Scottsdale, Arizona
  - Aclaris Investigational Site, Encino, California
  - Aclaris Investigational Site, Los Angeles, California
  - Aclaris Investigational Site, Tampa, Florida
  - Aclaris Investigational Site, Indianapolis, Indiana
  - Aclaris Investigational Site, Overland Park, Kansas
  - Aclaris Investigational Site, Omaha, Nebraska
  - Aclaris Investigational Site, Kew Gardens, New York
  - Aclaris Investigational Site, Newtown Square, Pennsylvania
  - Aclaris Investigational Site, Fountain Inn, South Carolina
  - Aclaris Investigational Site, Austin, Texas
  - Aclaris Investigational Site, San Antonio, Texas
  - Aclaris Investigational Site, Lynchburg, Virginia
  - Aclaris Investigational Site, Newport News, Virginia

REFERENCES:
- [Derived] Changelian P, Xu C, Mnich S, Hope H, Kostecki K, Hirsch J, Loh CY, Anderson D, Blinn J, Hockerman S, Dick E, Smith W, Monahan J, Raoof T, Forman S, Burt D, Barnes B, Gordon D, Walker N, Sudzina J, Tucker S, Jacobsen J. ATI-1777, a Topical Jak1/3 Inhibitor, May Benefit Atopic Dermatitis without Systemic Drug Exposure: Results from Preclinical Development and Phase 2a Randomized Control Study ATI-1777-AD-201. JID Innov. 2023 Nov 28;4(2):100251. doi: 10.1016/j.xjidi.2023.100251. eCollection 2024 Mar. PMID 38299059

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ATI-1777 | Vehicle
Started | 25 | 25
Received at Least 1 Dose of Study Drug | 23 | 25
Completed | 21 | 18
Not Completed | 4 | 7
Not completed — Adverse Event | 0 | 3
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Not Treated | 2 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | ATI-1777 | Vehicle | Total
Number analyzed (Participants) | 23 | 25 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (13.99) | 41.4 (14.31) | 42.3 (14.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 20 | 36
  Male | 7 | 5 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 15 | 12 | 27
  Black or African American | 7 | 10 | 17
  Asian | 1 | 0 | 1
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  Race missing | 0 | 1 | 1
  Multiple race | 0 | 1 | 1
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 18 | 20 | 38

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Score at Week 4
Description: The EASI evaluation was performed by the Principal Investigator and evaluated atopic dermatitis in each of 3 body regions (trunk [excluding groin and genitalia], upper extremities [excluding palms of hands], and lower extremities [excluding soles of feet]). The EASI scoring system uses a defined process to grade the severity of the signs of atopic dermatitis and the extent affected. EASI Scores ranged from 0-72, with higher scores indicative of more severe disease.
Time Frame: Baseline, Week 4
Population: Full Analysis Set: included all participants who were randomized and administered at least one dose of study medication. Data was imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | ATI-1777 | Vehicle
Number analyzed (Participants) | 23 | 25
percent change | -74.45 (6.455) | -41.43 (6.189)
Statistical Analysis 1: Comparison: ATI-1777 vs Vehicle; Test type: Superiority; p < 0.001, Mixed Model Repeated Measures (MMRM) — P-value is based on a 1-sided hypothesis test of the superiority of ATI-1777 relative to the vehicle. Significance level at α = 0.05; Least Square Means (LSM) % Differences = -33.01, 90% CI 2-sided [-47.95 to -18.08], Standard Error of Mean 8.971 — Fixed factors for treatment, visit, visit*treatment, baseline measurement. A compound symmetry covariance matrix was used to account for within-subject variability. Week 4: Least Square Means (LSM) % differences ATI-1777 arm minus vehicle arm

2. Secondary Outcome: Percent Change From Baseline in EASI Score at Days 8 and 15
Description: The EASI evaluation is performed by the Principal Investigator and will evaluate atopic dermatitis in each of 3 body regions (trunk [excluding groin and genitalia], upper extremities [excluding palms of hands], and lower extremities [excluding soles of feet]). The EASI scoring system uses a defined process to grade the severity of the signs of atopic dermatitis and the extent affected. EASI Scores range from 0-72, with higher scores indicative of more severe disease.
Time Frame: Baseline, Days 8 and 15
Population: Full Analysis Set: included all participants who were randomized and administered at least one dose of study medication. Data was imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | ATI-1777 | Vehicle
Number analyzed (Participants) | 23 | 25
percent change
  Day 8 | -35.95 (6.455) | -12.42 (6.189)
  Day 15 | -54.12 (6.455) | -30.68 (6.189)
Statistical Analysis 1: Comparison: ATI-1777 vs Vehicle; Day 8 statistical analysis; Test type: Superiority; p = 0.005, MMRM — [p-value comment as in outcome 1, analysis 1]; LSM % Differences = -23.53, 90% CI 2-sided [-38.47 to -8.59], Standard Error of Mean 8.971 — Fixed factors for treatment, visit, visit*treatment, baseline measurement. A compound symmetry covariance matrix was used to account for within-subject variability. Day 8: LSM % differences ATI-1777 arm minus vehicle arm
Statistical Analysis 2: Comparison: ATI-1777 vs Vehicle; Day 15 statistical analysis; Test type: Superiority; p = 0.005, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LSM % Differences = -23.44, 90% CI 2-sided [-38.38 to -8.50], Standard Error of Mean 8.971 — Fixed factors for treatment, visit, visit*treatment, baseline measurement. A compound symmetry covariance matrix was used to account for within-subject variability. Day 15: LSM % differences ATI-1777 arm minus vehicle arm

3. Secondary Outcome: Number of Participants Who Achieve 50% Improvement in EASI Score (EASI 50) by Week 4
Description: as for outcome 2
Time Frame: Week 4
Population: Full Analysis Set: included all participants who were randomized and administered at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-1777 | Vehicle
Number analyzed (Participants) | 23 | 25
Participants | 21 | 10
Statistical Analysis 1: Comparison: ATI-1777 vs Vehicle; Test type: Superiority; p < 0.001, Regression, Logistic — 1-sided p-value of responders in the treatment groups at 0.05 level of significance; Odds Ratio, log = 15.7, 90% CI 2-sided [3.9 to 63.2] — Active/Vehicle

4. Secondary Outcome: Number of Participants Who Achieve 75% Improvement in EASI Score (EASI-75) by Week 4
Description: as for outcome 2
Time Frame: Week 4
Population: Full Analysis Set: included all participants who were randomized and administered at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-1777 | Vehicle
Number analyzed (Participants) | 23 | 25
Participants | 15 | 6
Statistical Analysis 1: Comparison: ATI-1777 vs Vehicle; Test type: Superiority; p = 0.003, Regression, Linear — 1-sided p-value of responders in the treatment groups at 0.05 level of significance; Odds Ratio, log = 5.9, 90% CI 2-sided [2.1 to 17.0] — Active/Vehicle

5. Secondary Outcome: Number of Participants Who Achieve 90% Improvement in EASI Score (EASI-90) by Week 4
Description: as for outcome 2
Time Frame: Week 4
Population: Full Analysis Set: included all participants who were randomized and administered at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-1777 | Vehicle
Number analyzed (Participants) | 23 | 25
Participants | 7 | 5
Statistical Analysis 1: Comparison: ATI-1777 vs Vehicle; Test type: Superiority; p = 0.203, Regression, Logistic — 1-sided p-value of responders in the treatment groups at 0.05 level of significance; Odds Ratio, log = 1.7, 90% CI 2-sided [0.6 to 5.3] — Active/Vehicle

6. Secondary Outcome: Change From Baseline in Investigator Global Assessment (IGA) Score for Atopic Dermatitis at Days 8 and 15, and Week 4
Description: The IGA is a validated investigator's assessment of the average overall severity of participants' atopic dermatitis at a particular point in time. Scores ranged from 0-4, with higher scores indicative of more severe disease.
Time Frame: Baseline, Days 8 and 15, and Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATI-1777 | Vehicle
Number analyzed (Participants) | 23 | 25
units on a scale
  Day 8 | -0.50 (0.163) | -0.26 (0.156)
  Day 15 | -1.15 (0.163) | -0.66 (0.156)
  Week 4 | -1.59 (0.163) | -0.90 (0.156)
Statistical Analysis 1: Comparison: ATI-1777 vs Vehicle; Day 8 statistical analysis; Test type: Superiority; p = 0.148, MMRM — 1-sided p-value of responders in the treatment groups at 0.05 level of significance
Statistical Analysis 2: Comparison: ATI-1777 vs Vehicle; Day 15 statistical analysis; Test type: Superiority; p = 0.017, MMRM — 1-sided p-value of responders in the treatment groups at 0.05 level of significance
Statistical Analysis 3: Comparison: ATI-1777 vs Vehicle; Week 4 statistical analysis; Test type: Superiority; p = 0.002, MMRM — 1-sided p-value of responders in the treatment groups at 0.05 level of significance

7. Secondary Outcome: Change From Baseline in Percent of Body Surface Area (BSA) of Atopic Dermatitis at Days 8 and 15 and Week 4
Description: The total percentage of the participants BSA affected by atopic dermatitis was estimated by the investigator or designee using the handprint method, which estimates that the area of a participants' full handprint (fingers and thumbs together) constitutes 1% of their total BSA. Scores ranged from 0-100%, with higher scores indicative of increased percentage of atopic dermatitis on the skin.
Time Frame: Baseline, Days 8 and 15, and Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of BSA
Arm/Group | ATI-1777 | Vehicle
Number analyzed (Participants) | 23 | 25
percentage of BSA
  Day 8 | -1.55 (0.616) | -0.37 (0.590)
  Day 15 | -3.33 (0.616) | -1.57 (0.590)
  Week 4 | -5.59 (0.616) | -2.09 (0.590)
Statistical Analysis 1: Comparison: ATI-1777 vs Vehicle; Day 8 statistical analysis; Test type: Superiority; p = 0.088, MMRM — 1-sided p-value of responders in the treatment groups at 0.05 level of significance
Statistical Analysis 2: Comparison: ATI-1777 vs Vehicle; Day 15 statistical analysis; Test type: Superiority; p = 0.022, MMRM — 1-sided p-value of responders in the treatment groups at 0.05 level of significance
Statistical Analysis 3: Comparison: ATI-1777 vs Vehicle; Week 4 statistical analysis; Test type: Superiority; p < 0.001, MMRM — 1-sided p-value of responders in the treatment groups at 0.05 level of significance

8. Secondary Outcome: Change From Baseline in Peak Pruritus Numerical Rating Scale (PP-NRS) Score at Days 8 and 15, and Week 4
Description: The PP-NRS is a single patient-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours. Scores ranged from 0-10, with higher scores indicative of more severe itching.
Time Frame: Baseline, Days 8 and 15, and Week 4
Population: Full Analysis Set: included all participants who were randomized and administered at least one dose of study medication. Data was imputed using LOCF. Here, Overall Number of Participants Analyzed represents the participants evaluable for this measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATI-1777 | Vehicle
Number analyzed (Participants) | 23 | 24
units on a scale
  Day 8 | -2.18 (0.548) | -0.45 (0.536)
  Day 15 | -2.57 (0.548) | -1.41 (0.536)
  Week 4 | -2.92 (0.548) | -1.70 (0.536)
Statistical Analysis 1: Comparison: ATI-1777 vs Vehicle; Day 8 statistical analysis; Test type: Superiority; p = 0.014, MMRM — 1-sided p-value of responders in the treatment groups at 0.05 level of significance
Statistical Analysis 2: Comparison: ATI-1777 vs Vehicle; Day 15 statistical analysis; Test type: Superiority; p = 0.069, MMRM — 1-sided p-value of responders in the treatment groups at 0.05 level of significance
Statistical Analysis 3: Comparison: ATI-1777 vs Vehicle; Week 4 statistical analysis; Test type: Superiority; p = 0.060, MMRM — 1-sided p-value of responders in the treatment groups at 0.05 level of significance

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) through Day 42
Arm/Group | ATI-1777 | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/25
Other Adverse Events (participants affected / at risk) | 4/23 | 0/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ATI-1777 (N=23) | Vehicle (N=25)
Blood creatine phosphokinase increased (Blood and lymphatic system disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/69/NCT04598269/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/69/NCT04598269/SAP_001.pdf